CLINICAL TRIAL: NCT02981043
Title: Does "Aggressivity" of Endometriosis Correlate to Clinical History or Outcomes?
Acronym: Aggressivity
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Patrick Yeung Jr., MD, Principal Investigator, St. Louis University
Other Study IDs: 23924
Record Dates: First submitted 2016-10-04; First posted 2016-12-02 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood EDTA (about 10ml) (study related).
  2. Peritoneal tissue (about 3-4 samples each the size of 1 tsp) (SOC)
  3. Peritoneal fluid, if present (up to 100cc) (SOC) 4 Endometrial biopsy (1/4 to 1/2 inch long, (1/8 to 1/4 in width) (several SOC biopsies will be taken and one will be sent for research).
  5. Possibly small amount of ovarian tissue (if abnormal) (about size of 1 tsp) (SOC)
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical studies so far have been limited, and larger volume and multi-center studies studies are needed. The purpose of this pilot study is to look for a clinical correlations between the aggressivity panel developed from biomarkers thought to affect the progression or aggressivity of endometriosis, pain and quality of life.

Our goal with the study is find a correlation between the "aggressivity" of endometriosis with clinical factors determined in our study questionnaires. The "aggressivity panel" was pioneered by the EndoDiag lab in France, and was created using markers thought to affect the activity or progression of endometriosis. This information could lead to a better understanding of the disease, and ultimately lead to more targeted therapies.

If a patient returns for a second surgery we will ask their permission to use their slides from their first and seconed surgery to compare. The tissue that is being removed during the surgery as standard of care to make slides for the research study (there will not be an endometrial biopsy performed for research purposes with the second surgery). The slides from surgery 1 & surgery 2 will then be compared.

If a clinical correlation is found with the aggressivity panel, the goal would be to create a local lab and tissue bank here in the United States that could provide a basis for collaborative national (even international) research. Also, if a correlation is found, future investigation will look at correlations of the aggressivity panel and fertility outcomes. Results of this pilot study will help to direct studies of treatment protocols of the various stages of aggressivity of endometriosis.

DETAILED DESCRIPTION:
The study design is an investigator-initiated pilot, prospective cohort study (Canadian Task Force, II-3). Patients will not be randomized.

Consecutive subjects from age 14-55 will be recruited and included in the study if they are seeking treatment of pain and with suspected or known endometriosis. Patients who are menopausal (either chemically-induced, natural or surgical) will not be included in the study. Patients who are pregnant are not eligible for surgery, and not eligible to be in the study. Subjects will be excluded if they are found not to have endometriosis confirmed by histology. All surgeries are performed at a single institution, St. Mary's Hospital.

An ad hoc sample size calculation is not possible for this pilot study, since we have no historic data on which to base such a calculation. The goal is to acquire 45 panel results, as a reasonable amount of data for a pilot study, and given the funding available.

Quality of life (measured by the 100-point scale and by the EHP-5) and pain indices (measured by the VAS scale) will be measured at up to six different time points: before surgery, six months after surgery, and one year after each surgery. At each time point you will compare quality of life and each pain index across the four aggressivity groups of low, moderate, medium, and high using analysis of variance (ANOVA) or the non-parametric Kruskal-Wallis test depending on the normality of the distributions. Pairwise comparisons will also be made using independent students t test or the non-parametric Kolmogorov-Smirnov test depending on the normality of the distributions.

The follow-up time frame for each surgery will be 1 year. Patients will receive questionnaires pre op and at 6-months and 1 year for both the first surgery and the second surgery( if needed). The entire study will take about 4 years, including data analysis and publication. .

This study is related to IRB #20900. Subjects who consent to participate in this study may also be consented to participate in 20900. The pre-operative and follow-up questionnaires, and the standardized tools relating to QOL and depression are the same as in IRB#20900.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* 14-55 years of age
* Anyone seen at the Center for Endometriosis, including patients referred for the evaluation and management of pelvic pain
* Subjects must be having excision surgery for their endometriosis

Exclusion Criteria:

* Prior bilateral salpingo-oophorectomy, or post natural menopause
* Significant mental or chronic systemic illness that might confound pain assessment or the inability to complete the study.

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be identified, learn of the research and be recruited from the investigator's patient population.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Survey: "how aggressive the endometriosis might be" | At Surgery

IPD SHARING:
Plan to Share IPD: No